CLINICAL TRIAL: NCT06502535
Title: The Effects of Inulin and Inorganic Nitrate on Flow-Mediated Dilation and Gut Microbiome in Adults with Pre-Hypertension and Hypertension
Brief Title: Inulin and Nitrate's Effects on Vascular Health and Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 550689
Record Dates: First submitted 2024-05-14; First posted 2024-07-16 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Endothelial Dysfunction; High Blood Pressure; Gut Microbiota Dysbiosis and Nutrition
MeSH Terms: conditions — Hypertension | interventions — Inulin; potassium nitrate

STUDY DESIGN:
Intervention Model Description: Participants will be assigned randomly to receive either A) a combination of inulin and nitrate, or B) inulin alone. This will be done following a crossover and counterbalanced design, ensuring that all participants will receive both treatments in a randomised order.
Who Masked: Participant, Investigator
Masking Description: This study will be conducted under a double-blind setup, which implies that neither the participants nor the researcher will be aware of whether the participants are being given inulin or a combination of inulin and nitrate. The supplements will be labelled A and B by an independent party otherwise not involved in the study, and the investigator and participants will not know which supplement is which letter during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inulin (15 g) (Experimental): Participants will receive 15 g inulin in powder form once daily for 4 weeks.
  Interventions: Dietary Supplement: Inulin
- Inulin (15 g) and potassium nitrate (1300 mg) (Experimental): Participants will receive 15 g inulin in powder form once daily for 4 weeks and 1300 mg potassium nitrate in powder form once daily for 4 weeks.
  Interventions: Dietary Supplement: Potassium nitrate and inulin

INTERVENTIONS:
Dietary Supplement: Inulin — 15 g inulin once daily for 4 weeks.
  Arms: Inulin (15 g)
Dietary Supplement: Potassium nitrate and inulin — 1300 mg potassium nitrate once daily for 4 weeks and 15 g inulin once daily for 4 weeks.
  Arms: Inulin (15 g) and potassium nitrate (1300 mg)

SUMMARY:
Previous research has revealed that adults with pre-hypertensive and hypertensive blood pressure levels typically exhibit impaired vasodilation, which is a crucial aspect of blood vessel function, due to decreased nitric oxide production. Flow-mediated dilation (FMD) is a widely used technique for assessing vasodilation, which gauges the capacity of blood vessels to widen in response to increased blood flow. Nitrate supplements have been shown to enhance blood vessel function both in the short and long term by elevating nitric oxide (NO) production. Similarly, acetate, a by-product of fibre digestion, has demonstrated anti-inflammatory effects in the gut and may also increase NO production. However, further investigation is needed to determine whether these two supplements work synergistically to improve FMD responses by augmenting NO production in the human body. This study will involve administering inulin plus nitrate supplements to adults aged 45-74 with untreated high blood pressure (120-139/80-89 mmHg and 140/90 mmHg or higher) for a period of 4 weeks, followed by a subsequent 4-week period where only inulin supplements are consumed. The supplements will be provided in the form of powder, to be mixed with water, and will be given in a cross-over and counterbalanced order. Various measurements, including brachial artery function, faecal samples, blood pressure, plasma nitrate and nitrite levels, plasma short-chain fatty acid levels, red blood cell and whole blood S-Nitrosothiols, and salivary nitrate and nitrite levels, will be taken at the baseline and after each supplementation period. Additionally, acute supplementation measurements will be collected on two separate occasions before the start of the longer-term supplement regimen.

DETAILED DESCRIPTION:
Endothelial dysfunction contributes to the increased cardiovascular risk associated with high blood pressure levels (e.g., 120-139/80-89 mmHg and 140/90 mmHg or higher), and it is considered as an early event in the development of atherosclerotic vascular disease. Mechanistically, endothelial dysfunction is characterised by a reduced bioavailability of the endothelium-derived molecule nitric oxide (NO), which is reflected by impaired brachial artery flow-mediated dilation (FMD). However, endothelial dysfunction is largely preventable by its early detection, thus approaches that might restore the loss of NO in the body could have obvious therapeutic potential.

Consumption of the prebiotic fibre inulin has been shown to increase the fermentation of bacterial-derived metabolites such as acetate by our gut microbiome. While increased acetate has local benefits in the gut (i.e., anti-inflammatory, lower luminal pH), it also has the potential to improve endothelial health. Research has shown that acetate can increase NO bioavailability via the activation of the NO synthase pathway by increasing phosphorylation of endothelial NO synthase (eNOS), a key enzyme in the maintenance of endothelial homeostasis, following a 15-day supplementation with inulin. Similarly, NO is produced following the consumption of nitrate, with individual responses being dependent on the basal eNOS activity. Therefore, individuals with compromised eNOS activity (e.g., pre- and hypertensive) might show an augmented response to nitrate supplementation. Since both nitrate and inulin supplementations can increase NO production, it is possible that their combined ingestion might enhance endothelial function to a greater extent. When supplemented in isolation, nitrate proved an effective dietary strategy to ameliorate endothelial dysfunction in older and clinical populations. For example, a 4-week chronic dietary nitrate supplementation (400 mg nitrate/day) was associated with an increased peak brachial artery FMD of 1.0% (95% CI, 0.3-1.5; p < 0.001), which was not evident in the placebo group. Similarly, following a 4-week dietary nitrate supplementation (400 mg nitrate/day), brachial artery FMD (%) values increased significantly in the nitrate group compared to the placebo group. Unlike nitrate, the effects of inulin on brachial artery FMD in humans are yet to be established. Preliminary findings demonstrated an enhancement of endothelial function after inulin supplementation in mice. These findings were further supported by another study which demonstrated a brachial artery FMD increase of ~1% following a 3-month prebiotic supplementation with 12 g fructo-oligosaccharides in clinical patients with less severe endothelial dysfunction.

To date, no studies that the investigators are aware of have explored the role of nitrate and inulin in combination; however, based on the above, these two nutrients have the potential to work synergistically. Therefore, the primary aim of this study is to assess whether adding nitrate to inulin during a 4-week chronic supplementation might lead to an increase in brachial artery FMD in middle-aged and youngest elderly adults (45-74 years old) with elevated blood pressure and compare this response to inulin supplemented in isolation. The secondary aims of this study include brachial artery FMD % changes at 4 h post-consumption of a single dose of 15 g inulin and 1300 mg potassium nitrate combined and 15 g inulin supplemented in isolation. This study will also explore whether changes in brachial artery FMD % following the two supplementations are mediated by potential changes in the gut microbiome composition and diversity that may occur following prebiotics supplementation. Further secondary outcomes of the study will investigate differences in plasma nitrate, nitrite, and short-chain fatty acids (SCFAs) following both types of supplementation. Additionally, the study will examine changes in the levels of S-nitrosothiols (RSNO) in red blood cells and whole blood. The study will also compare changes in resting blood pressure between the combined inulin and nitrate supplementation and the inulin-only supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Adults aged 45-74
* Adults with untreated elevated blood pressure as SBP 120 to 129 mm Hg and DBP < 80 mm Hg or untreated stage 1 hypertension (i.e., pre-hypertension) as SBP 130 to 139 mm Hg or DBP 80 to 89 mm Hg or untreated stage 2 hypertension as SBP equal to or higher than 140 mm Hg or DBP equal to or higher than 90 mm Hg (ACC/AHA and ESC/ESH guidelines and Blood Pressure UK)
* Weight-stable in the 3 months prior to enrolment (self-report)

Exclusion Criteria:

* Body mass index > 40 kg/m^2 at screening;
* History of symptomatic coronary artery disease, stroke, or other known atherosclerotic disease;
* History of gastrointestinal disease (e.g., irritable bowel syndrome, inflammatory bowel disease, coeliac disease, Chron's disease) or former abdominal surgery, weight loss surgery e.g., gastric by-pass (except for appendectomy);
* History of chronic viral hepatitis (including presence of hepatitis B surface antigen or hepatitis C antibody), or other chronic hepatic disorders;
* History of malignancy within the past 5 years, other than non-melanoma skin cancer;
* History of diabetes and/or any endocrine disorder;
* Current use of nitrate medications, including glyceryl trinitrate (GTN), isosorbide dinitrate and isosorbide mononitrate and blood pressure medications;
* Consumption of a low calorie or other special diet during the last month prior to the study, or if following a slimming or medically prescribed diet, or a vegan or macrobiotic lifestyle;
* Use of antibiotics during the three months prior to screening;
* Consumption of pre- or probiotics during the last month prior to screening and during the study, unless discontinued 3 weeks before the start of the trial. This is referred to the use of supplements only and NOT foods containing probiotics and/or prebiotics foods;
* Consumption of dietary supplements such as vitamins C and E during the last month prior to the screening and during the trial, unless discontinued 3 weeks before the start of the trial;
* Consumption of fish oil 6 weeks prior to the screening and during the trial, unless discontinued 6 weeks before the start of the trial;
* Allergies or intolerance against the substances used in the study and/or food intolerances associated with gastrointestinal upset;
* Any apparent dependence on or abuse of alcohol, tobacco, and cannabis products;
* Pregnancy, breast-feeding, or plans to become pregnant during the duration of the study;
* Current use of nitrate supplements in the form of beetroot juice, beetroot crystals, potassium nitrate and sodium nitrate, including L-arginine or L-citrulline supplements.
* Self-reported use of antimicrobial mouthwash or tongue scrapes, unless discontinued during the trial.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation (FMD) with ultrasound to detect a change in brachial artery FMD | Day 0, Month 3
  Absolute percentage change in FMD response between the 'inulin plus nitrate' and 'inulin' supplementations, measured from baseline to the 4-week chronic supplementation.
Plasma nitrite and nitrate levels | Day 0, Month 3
  Differences in the concentrations of plasma nitrate and nitrite between the 'inulin plus nitrate' and 'inulin' supplementations as assessed by chemiluminescence, measured from baseline to the 4-week chronic supplementation.
Plasma Short-Chain Fatty Acid (SCFA) levels | Day 0, Month 3
  Differences in the concentrations of plasma acetate, butyrate, and propionate between the 'inulin plus nitrate' and 'inulin' supplementations as assessed by liquid chromatography coupled with tandem mass spectrometry, measured from baseline to the 4-week chronic supplementation.
Gut microbial composition using 16S sequencing | Day 0, Month 3
  Changes in microbial composition, including alpha and beta diversity indexes, will be evaluated using the 16S rRNA V3-V4 region. These changes will be observed from baseline to the 4-week intervention following both inulin plus nitrate and inulin-only supplementation.
Gut microbial composition using 16S sequencing | Day 0, Month 3
  Changes in microbial composition, including Least Discriminant Analysis (LDA) evaluated using the 16S rRNA V3-V4 region, will be observed from baseline to the end of the 4-week intervention following supplementation with inulin plus nitrate and inulin alone.
Gut microbial composition using 16S sequencing | Day 0, Month 3
  Changes in microbial composition, including the relative abundances of Operational Taxonomic Units (OTUs), will be evaluated using the 16S rRNA V3-V4 region. These changes will be observed from baseline to the end of the 4-week intervention following supplementation with inulin plus nitrate and inulin alone.

SECONDARY OUTCOMES:
Flow-mediated dilation (FMD) with ultrasound to detect a change in brachial artery FMD | Baseline, 4 hour post supplement consumption
  Absolute percentage change in FMD response between the 'inulin plus nitrate' and 'inulin' supplementations, measured from baseline to 4 h post-consumption of the supplements.
Plasma nitrite and nitrate levels | Baseline, 4 hour post supplement consumption
  Differences in the concentrations of plasma nitrate and nitrite between the 'inulin plus nitrate' and 'inulin' supplementations as assessed by chemiluminescence, measured from baseline to 4 h post-consumption of the supplements.
Plasma Short-Chain Fatty Acid (SCFA) levels | Baseline, 4 hour post supplement consumption
  Differences in the concentrations of plasma acetate, butyrate, and propionate between the 'inulin plus nitrate' and 'inulin' supplementations as assessed by liquid chromatography coupled with tandem mass spectrometry, measured from baseline to 4 h post-consumption of the supplements.
S-nitrosothiols (RSNO) in red blood cells and whole blood | Baseline, 4 hour post supplement consumption
  Differences in the concentrations of RSNO in red blood cells and whole blood following the 'inulin plus nitrate' and 'inulin' supplementations as assessed from chemiluminescence, measured from baseline to 4 h post-consumption of the supplements.
S-nitrosothiols (RSNO) in red blood cells and whole blood | Day 0, Month 3
  Differences in the concentrations of RSNO in red blood cells and whole blood following the 'inulin plus nitrate' and 'inulin' supplementations as assessed from chemiluminescence, measured from baseline to the 4-week intervention.
Resting blood pressure | Baseline, 4 hour post supplement consumption
  Differences in resting blood pressure following the 'inulin plus nitrate' and the 'inulin' supplementations as assessed by an automatic sphygmomanometer, measured from baseline to 4 h post-consumption of the supplements.
Resting blood pressure | Day 0, Month 3
  Differences in resting blood pressure following the 'inulin plus nitrate' and the 'inulin' supplementations as assessed by an automatic sphygmomanometer, measured from baseline to the 4-week intervention.
Tolerability of inulin defined by gastrointestinal wellbeing | Day 0, Month 3
  Tolerability of a 4-week intervention with inulin with or without nitrate, assessed by completion of gastrointestinal wellbeing questionnaires, also known as the Gastrointestinal Symptom Rating Scale (GSRS). GSRS score will be calculated as per Revicki 1997:
  Response scale
  1. No discomfort at all
  2. Slight discomfort
  3. Mild discomfort
  4. Moderate discomfort
  5. Moderately severe discomfort
  6. Severe discomfort
  7. Very severe discomfort
  The 14 items combine into five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation.
Rate of habitual fibre intake before and during the intervention | Pre intervention, at baseline
  Participants will be categorised based on their habitual dietary fibre intake to determine if the effects of the supplemented inulin are independent of their overall fibre consumption.
  The questionnaire includes 5 questions addressing the intake from the five main food groups contributing to fibre intake: fruit, vegetables, bread and cereals, nuts and seeds, and legumes. The intake of these food groups will be evaluated using the following scale:
  Never Less than 1 serving per month 1-3 servings per month
  1 serving per week 2-4 servings per week 5-6 servings per week
  1. serving per day
  2. servings per day
  3. servings per day
  4. servings per day
  5. servings per day
  6. or more servings per day
Dietary intake | Day 0, Month 3
  4-day recall questionnaire filled out during 4 different occasions to evaluate dietary intake, including macronutrients and caloric intake.
Body weight | Day 0, Month 3
  Changes in body weight in Kg following supplementation with 'inulin plus nitrate' and 'inulin' will be measured with the use of electronic scales.
Body fat percentage | Day 0, Month 3
  Changes in body fat percentage following supplementation with 'inulin plus nitrate' and 'inulin' will be assessed using bioimpedance analysis.
Hip circumference | Day 0, Month 3
  The changes in hip circumference, measured at the largest circumference around the buttocks, following supplementation with 'inulin plus nitrate' and 'inulin,' will be used to calculate the waist-to-hip ratio in conjunction with waist measurement, from baseline to the 4-week intervention.
Waist circumference | Day 0, Month 3
  The changes in waist circumference, measured halfway between the lower ribs and the iliac crest, following supplementation with 'inulin plus nitrate' and 'inulin', will be used to calculate the waist-to-hip ratio in conjunction with hip measurement, from baseline to the 4-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Torquati, PhD, Principal Investigator — University of Exeter; Jessica Virgili, MSc, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armani RG, Carvalho AB, Ramos CI, Hong V, Bortolotto LA, Cassiolato JL, Oliveira NF, Cieslarova Z, do Lago CL, Klassen A, Cuppari L, Raj DS, Canziani MEF. Effect of fructooligosaccharide on endothelial function in CKD patients: a randomized controlled trial. Nephrol Dial Transplant. 2021 Dec 31;37(1):85-91. doi: 10.1093/ndt/gfaa335. PMID 33411910
- [Background] Bhardwaj R, Dod H, Sandhu MS, Bedi R, Dod S, Konat G, Chopra HK, Sharma R, Jain AC, Nanda N. Acute effects of diets rich in almonds and walnuts on endothelial function. Indian Heart J. 2018 Jul-Aug;70(4):497-501. doi: 10.1016/j.ihj.2018.01.030. Epub 2018 Feb 1. PMID 30170643
- [Background] Boets E, Deroover L, Houben E, Vermeulen K, Gomand SV, Delcour JA, Verbeke K. Quantification of in Vivo Colonic Short Chain Fatty Acid Production from Inulin. Nutrients. 2015 Oct 28;7(11):8916-29. doi: 10.3390/nu7115440. PMID 26516911
- [Background] Carlstrom M, Liu M, Yang T, Zollbrecht C, Huang L, Peleli M, Borniquel S, Kishikawa H, Hezel M, Persson AE, Weitzberg E, Lundberg JO. Cross-talk Between Nitrate-Nitrite-NO and NO Synthase Pathways in Control of Vascular NO Homeostasis. Antioxid Redox Signal. 2015 Aug 1;23(4):295-306. doi: 10.1089/ars.2013.5481. Epub 2014 Feb 6. PMID 24224525
- [Background] Catry E, Bindels LB, Tailleux A, Lestavel S, Neyrinck AM, Goossens JF, Lobysheva I, Plovier H, Essaghir A, Demoulin JB, Bouzin C, Pachikian BD, Cani PD, Staels B, Dessy C, Delzenne NM. Targeting the gut microbiota with inulin-type fructans: preclinical demonstration of a novel approach in the management of endothelial dysfunction. Gut. 2018 Feb;67(2):271-283. doi: 10.1136/gutjnl-2016-313316. Epub 2017 Apr 4. PMID 28377388
- [Background] Craighead DH, Freeberg KA, Seals DR. Vascular Endothelial Function in Midlife/Older Adults Classified According to 2017 American College of Cardiology/American Heart Association Blood Pressure Guidelines. J Am Heart Assoc. 2020 Sep;9(17):e016625. doi: 10.1161/JAHA.120.016625. Epub 2020 Aug 20. PMID 32815446
- [Background] Heiss C, Rodriguez-Mateos A, Kelm M. Central role of eNOS in the maintenance of endothelial homeostasis. Antioxid Redox Signal. 2015 May 10;22(14):1230-42. doi: 10.1089/ars.2014.6158. Epub 2014 Dec 10. PMID 25330054
- [Background] Inaba Y, Chen JA, Bergmann SR. Prediction of future cardiovascular outcomes by flow-mediated vasodilatation of brachial artery: a meta-analysis. Int J Cardiovasc Imaging. 2010 Aug;26(6):631-40. doi: 10.1007/s10554-010-9616-1. Epub 2010 Mar 26. PMID 20339920
- [Background] Jones T, Dunn EL, Macdonald JH, Kubis HP, McMahon N, Sandoo A. The Effects of Beetroot Juice on Blood Pressure, Microvascular Function and Large-Vessel Endothelial Function: A Randomized, Double-Blind, Placebo-Controlled Pilot Study in Healthy Older Adults. Nutrients. 2019 Aug 2;11(8):1792. doi: 10.3390/nu11081792. PMID 31382524
- [Background] Kapil V, Khambata RS, Robertson A, Caulfield MJ, Ahluwalia A. Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study. Hypertension. 2015 Feb;65(2):320-7. doi: 10.1161/HYPERTENSIONAHA.114.04675. Epub 2014 Nov 24. PMID 25421976
- [Background] Kleinbongard P, Dejam A, Lauer T, Jax T, Kerber S, Gharini P, Balzer J, Zotz RB, Scharf RE, Willers R, Schechter AN, Feelisch M, Kelm M. Plasma nitrite concentrations reflect the degree of endothelial dysfunction in humans. Free Radic Biol Med. 2006 Jan 15;40(2):295-302. doi: 10.1016/j.freeradbiomed.2005.08.025. Epub 2005 Nov 10. PMID 16413411
- [Background] Koch CD, Gladwin MT, Freeman BA, Lundberg JO, Weitzberg E, Morris A. Enterosalivary nitrate metabolism and the microbiome: Intersection of microbial metabolism, nitric oxide and diet in cardiac and pulmonary vascular health. Free Radic Biol Med. 2017 Apr;105:48-67. doi: 10.1016/j.freeradbiomed.2016.12.015. Epub 2016 Dec 16. PMID 27989792
- [Background] Medina-Leyte DJ, Zepeda-Garcia O, Dominguez-Perez M, Gonzalez-Garrido A, Villarreal-Molina T, Jacobo-Albavera L. Endothelial Dysfunction, Inflammation and Coronary Artery Disease: Potential Biomarkers and Promising Therapeutical Approaches. Int J Mol Sci. 2021 Apr 8;22(8):3850. doi: 10.3390/ijms22083850. PMID 33917744
- [Background] Park KH, Park WJ. Endothelial Dysfunction: Clinical Implications in Cardiovascular Disease and Therapeutic Approaches. J Korean Med Sci. 2015 Sep;30(9):1213-25. doi: 10.3346/jkms.2015.30.9.1213. Epub 2015 Aug 13. PMID 26339159
- [Background] Rios-Covian D, Ruas-Madiedo P, Margolles A, Gueimonde M, de Los Reyes-Gavilan CG, Salazar N. Intestinal Short Chain Fatty Acids and their Link with Diet and Human Health. Front Microbiol. 2016 Feb 17;7:185. doi: 10.3389/fmicb.2016.00185. eCollection 2016. PMID 26925050
- [Background] Velmurugan S, Gan JM, Rathod KS, Khambata RS, Ghosh SM, Hartley A, Van Eijl S, Sagi-Kiss V, Chowdhury TA, Curtis M, Kuhnle GG, Wade WG, Ahluwalia A. Dietary nitrate improves vascular function in patients with hypercholesterolemia: a randomized, double-blind, placebo-controlled study. Am J Clin Nutr. 2016 Jan;103(1):25-38. doi: 10.3945/ajcn.115.116244. Epub 2015 Nov 25. PMID 26607938